CLINICAL TRIAL: NCT03534895
Title: Does the Preoperative Midazolam Dose Affect Postoperative Pain? - a Multicentric Randomized Controlled Trial in Ambulatory Surgery
Brief Title: Does the Preoperative Midazolam Dose Affect Postoperative Pain?
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidade do Porto (Other)
Collaborators: Centro Hospitalar de Entre o Douro e Vouga (Other); Centro Hospitalar de Vila Nova de Gaia/Espinho (Other)
Responsible Party: Principal Investigator, Caroline Dahlem, Principal Investigator, Universidade do Porto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Midazolam RCT
Record Dates: First submitted 2018-04-22; First posted 2018-05-23 (Actual); Last update posted 2018-05-23 (Actual); Status verified 2018-05

CONDITIONS: Pain, Postoperative
Keywords: midazolam; ambulatory surgery
MeSH Terms: conditions — Pain, Postoperative | interventions — Midazolam; Saline Solution; Anesthesia, Spinal; Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- PC1 (Placebo Comparator): 5mL normal saline intravenous, single-administration, as pre-medication
  Interventions: Other: Normal saline; Procedure: Spinal anesthesia; Procedure: Surgery; Drug: Postoperative analgesia; Drug: Rescue analgesia; Drug: Wound infiltration; Drug: Analgesia at home
- PC2 (Experimental): midazolam 0.02mg/Kg in 5mL normal saline, intravenous, single-administration, as pre-medication
  Interventions: Drug: Midazolam Injectable Solution; Other: Normal saline; Procedure: Spinal anesthesia; Procedure: Surgery; Drug: Postoperative analgesia; Drug: Rescue analgesia; Drug: Wound infiltration; Drug: Analgesia at home
- PC3 (Experimental): midazolam 0.06mg/Kg in 5mL normal saline, intravenous, single-administration, as pre-medication
  Interventions: Drug: Midazolam Injectable Solution; Other: Normal saline; Procedure: Spinal anesthesia; Procedure: Surgery; Drug: Postoperative analgesia; Drug: Rescue analgesia; Drug: Wound infiltration; Drug: Analgesia at home

INTERVENTIONS:
Drug: Midazolam Injectable Solution — intravenous
  Other Names: Dormicum
  Arms: PC2; PC3
Other: Normal saline — intravenous
Procedure: Spinal anesthesia — 8mg of heavy bupivacaine 0.5% injected in the subarachnoid space, during lateral decubitus
Procedure: Surgery — Open inguinal hernia repair, varicose vein stripping, knee arthroscopy or hallux valgus surgery
Drug: Postoperative analgesia — IV acetaminophen 1g + IV ketorolac 30mg
Drug: Rescue analgesia — Tramadol 2mg/Kg IV in 100mL of normal saline, if pain NRS>3.
Drug: Wound infiltration — Wound infiltration with 10mL of ropivacaine 0.75%, in open inguinal hernia repair
Drug: Analgesia at home — Oral acetaminophen 1g 6/6h + ibuprofen 400mg 8/8h (+ rescue analgesia with tramadol 50mg 6/6h)

SUMMARY:
To investigate whether midazolam has any effect on postoperative pain in outpatient surgery, the investigators will assess the impact of different midazolam doses on pain scores 24h, 7 days and 3 months after ambulatory surgery.

The investigators hypothesize that patients being administered higher midazolam doses will refer more pain.

DETAILED DESCRIPTION:
Systemic midazolam prescribed perioperatively might have impact on pain, with studies suggesting antinociceptive and hyperalgesic effects. Anxiety might be a confounder in this association. In order to investigate the effect of midazolam on postoperative pain, a clinical trial will be conducted in Portuguese ambulatory surgery units. A convenience sample with consecutive design will include patients admitted for open inguinal hernia repair, varicose vein stripping, knee arthroscopy or hallux valgus surgery under spinal anesthesia. Patients will be randomized into 3 premedication groups, and this randomization will be stratified for each centre and each type of surgery. Postoperative pain will be blindly assessed by telephone interviews at 24h, 7 days, and 3 months.

The investigators will use multiple regression models to explore the interaction of midazolam dose with preoperative anxiety, gender and chronic benzodiazepine use, as they hypothesize there might be a differential effect of midazolam on postoperative pain amongst these subgroups.

ELIGIBILITY:
Inclusion Criteria:

* adult patients submitted to open inguinal hernia repair, varicose vein stripping, knee arthroscopy or hallux valgus surgery in Portuguese ambulatory surgery units

Exclusion Criteria:

* psychiatric disorders
* alcoholism
* illiteracy or poor understanding of Portuguese language
* history of chronic pain under opioids
* recurrent surgery
* contraindication for midazolam or deep sedation
* contraindication for spinal anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2019-05 (Estimated); Primary Completion 2020-05 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain | Day 1 after surgery
  Assessed by the Brief Pain Inventory severity score (24h recall time): mean of 4 items assessing pain at the moment of the interview, on average, at its least and at its worst during the last 24h

SECONDARY OUTCOMES:
Postoperative pain | Day 7 after surgery
  Assessed by the Brief Pain Inventory severity score (24h recall time): mean of 4 items assessing pain at the moment of the interview, on average, at its least and at its worst during the last 24h. Features of neuropathic pain as assessed by DN4 patient-reported symptoms
Postoperative pain | Month 3 after surgery
  Assessed by the Brief Pain Inventory severity score (24h recall time): mean of 4 items assessing pain at the moment of the interview, on average, at its least and at its worst during the last 24h. Features of neuropathic pain as assessed by DN4 patient-reported symptoms
Pain interference in daily life | Day 1 after surgery
  Assessed by the Brief Pain Inventory interference score (24h recall time): interference of pain in general activity, mood, walking ability, normal work, relations with other people, sleep and enjoyment of life.
Pain interference in daily life | Day 7 after surgery
  Assessed by the Brief Pain Inventory interference score (24h recall time): interference of pain in general activity, mood, walking ability, normal work, relations with other people, sleep and enjoyment of life.
Pain interference in daily life | Month 3 after surgery
  Assessed by the Brief Pain Inventory interference score (24h recall time): interference of pain in general activity, mood, walking ability, normal work, relations with other people, sleep and enjoyment of life.
Analgesic consumption | Day 1 after surgery
  Total analgesic drugs taken in a time period (first day after surgery)
Analgesic consumption | Day 7 after surgery
  Total analgesic drugs taken in a time period (first week after surgery)
Patient satisfaction | Day 7 after surgery
  NRS 0-10
Patient satisfaction | Month 3 after surgery
  NRS 0-10
Adverse events | Day 7 after surgery
  Number of patients with adverse events like bleeding, nausea, uncontrolled pain
Global surgery recovery index | Month 3 after surgery
  Global surgery recovery index (0-100%)

CONTACTS AND LOCATIONS:
Locations (2):
- Portugal (2):
  - Centro Hospitalar Entre Douro e Vouga, EPE, Santa Maria da Feira
  - Centro Hospitalar Vila Nova de Gaia / Espinho, EPE, Vila Nova de Gaia

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article might be shared with other researchers after deidentification.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 6 months following article publication.
Access Criteria: Proposals should be directed to caroline.dahlem@gmail.com. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Background] Mantegazza P, Parenti M, Tammiso R, Vita P, Zambotti F, Zonta N. Modification of the antinociceptive effect of morphine by centrally administered diazepam and midazolam. Br J Pharmacol. 1982 Apr;75(4):569-72. doi: 10.1111/j.1476-5381.1982.tb09175.x. PMID 6121598
- [Background] Tatsuo MA, Salgado JV, Yokoro CM, Duarte ID, Francischi JN. Midazolam-induced hyperalgesia in rats: modulation via GABA(A) receptors at supraspinal level. Eur J Pharmacol. 1999 Apr 1;370(1):9-15. doi: 10.1016/s0014-2999(99)00096-5. PMID 10323274
- [Background] Frolich MA, Zhang K, Ness TJ. Effect of sedation on pain perception. Anesthesiology. 2013 Mar;118(3):611-21. doi: 10.1097/ALN.0b013e318281592d. PMID 23314164
- [Background] Kain ZN, Sevarino F, Pincus S, Alexander GM, Wang SM, Ayoub C, Kosarussavadi B. Attenuation of the preoperative stress response with midazolam: effects on postoperative outcomes. Anesthesiology. 2000 Jul;93(1):141-7. doi: 10.1097/00000542-200007000-00024. PMID 10861157
- [Background] Day MA, Rich MA, Thorn BE, Berbaum ML, Mangieri EA. A placebo-controlled trial of midazolam as an adjunct to morphine patient-controlled analgesia after spinal surgery. J Clin Anesth. 2014 Jun;26(4):300-8. doi: 10.1016/j.jclinane.2013.12.011. Epub 2014 Jun 2. PMID 24882605
- [Background] Okulicz-Kozaryn I, Kaminska E, Luczak J, Szczawinska K, Kotlinska-Lemieszek A, Baczyk E, Mikolajczak P. The effects of midazolam and morphine on analgesic and sedative activity of ketamine in rats. J Basic Clin Physiol Pharmacol. 2000;11(2):109-25. doi: 10.1515/jbcpp.2000.11.2.109. PMID 11037766
- [Background] Hasani A, Maloku H, Sallahu F, Gashi V, Ozgen SU. Preemptive analgesia with midazolam and diclofenac for hernia repair pain. Hernia. 2011 Jun;15(3):267-72. doi: 10.1007/s10029-010-0772-y. Epub 2010 Dec 28. PMID 21188440